CLINICAL TRIAL: NCT07217132
Title: Monitoring the Use of Collagen Dura Membrane - Suturable (DMS) in the Post-market Phase
Brief Title: Clinical Investigation Plan - Post-market Clinical Follow-up Study Collagen Dura Membrane - Suturable
Status: Not yet recruiting | Type: Observational
Sponsor: Collagen Matrix (Industry)
Collaborators: Baptist Health South Florida (Other)
Responsible Party: Sponsor
Other Study IDs: CIP.033.2
Record Dates: First submitted 2025-10-13; First posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Repair of Dura Mater

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Post-market Study — Prospective case series without a concurrent comparator group.

SUMMARY:
Monitoring the use of Collagen Dura Membrane - Suturable (DMS) in the post-market phase

DETAILED DESCRIPTION:
A prospective, post-market clinical study at a maximum of three sites, with an enrollment of 54 subjects. The primary endpoint of the study will be the rate of adverse events related to the Subject Device requiring surgical intervention. The date of each event will be recorded and assessed, including at least one timepoint of 9 months of more post-operatively. Secondary endpoints will include all adverse events (i.e., infection, CSF Leak, and Pseudomeningocele), score of adequacy of product performance, score for product handling at implantation, and score for product adaptability at implantation.

No original patient records or patient identifying information will be disclosed to Collagen Matrix.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a dural defect requiring repair with a dural substitute
* Patient is 18 years or older
* Patient of child-bearing potential is not pregnant or nursing

Exclusion Criteria:

* Patients with a known history of hypersensitivity to bovine derived materials
* Patients that are non-English speaking
* Subjects requiring Legally Authorized Representative

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The general population will be included in the study where a dura substitute is required for the repair of dura mater.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Rate of Adverse Events Requiring Surgical Intervention | 9 months
  Rate of adverse events related to subject device and requiring surgical intervention.

SECONDARY OUTCOMES:
Rate of Adverse Events | 9 months
  Rate of all product related adverse events or complications.
Score of adequacy of product performance | 9 months
  rated yes/no by clinician
Score for Product Handling at Implantation | 9 months
  Rated on a scale from 1 (poor) to 4 (excellent) by clinician.
Score for Product Adaptability at Implantation | 9 months
  Rate on a scale of 1 (poor) to 4 (excellent) by clinician.

CONTACTS AND LOCATIONS:
Locations (1):
- Baptist Health South Florida, Miami, Florida, United States